CLINICAL TRIAL: NCT02704806
Title: Immunologic Analysis of Aspired Thromb and Circulatory Immune Cell in AMI Patients
Brief Title: Immunologic Analysis of Peripheral Blood and Aspirated Thromb In AMI Patients
Acronym: ATAIA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Mingyou Zhang, attending physician, Jilin University
Other Study IDs: Cthromb20160401
Record Dates: First submitted 2016-03-05; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Immunol Feature in Circulation and Thromb in AMI Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Thromb will be abtained with aspiration device during PCI intervention, peripheral blood will be abtained as well for study.
Oversight: Data Monitoring Committee: No

SUMMARY:
Researchers use FCM to analyze the immunol cell feature and its corresponding activation status, as well as the thromb aspirated through the thromb aspiration device in AMI patients

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated AMI patients

Exclusion Criteria:

* any self immune disease and recent (within 1 month) or any chronic infection

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute myocardial infarction patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
immunologic feature of AMI patients | 1 month